CLINICAL TRIAL: NCT00545480
Title: A Randomized, Open-label Study to Investigate the Impact of Bone Marker Feedback on Persistence to Once Monthly Oral Bonviva (Ibandronate) Treatment for Post-menopausal Osteoporosis.
Brief Title: SUMMIT Study: A Study of Persistence to Bonviva (Ibandronate) Once Monthly in Women With Post-Menopausal Osteoporosis.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML19358
Record Dates: First submitted 2007-10-16; First posted 2007-10-17 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-08

CONDITIONS: Post Menopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Ibandronic Acid

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: ibandronate [Bonviva/Boniva]
- 2 (Active Comparator)
  Interventions: Drug: ibandronate [Bonviva/Boniva]

INTERVENTIONS:
Drug: ibandronate [Bonviva/Boniva] — 150mg po monthly for 12 months (with feedback)
  Arms: 1
Drug: ibandronate [Bonviva/Boniva] — 150mg po monthly for 12 months (without feedback)
  Arms: 2

SUMMARY:
This 2 arm study will assess the impact of bone marker feedback, using blood sampling and communication of results at week 5, on persistence to monthly Bonviva (150mg po) in women with post-menopausal osteoporosis. The study will also assess safety, quality of life and patient satisfaction. All patients will receive Bonviva 150mg po monthly, and will be randomized into the bio-feedback or no bio-feedback study arms. The anticipated time on study treatment is 3-12 months, and the target sample size is 500+ individuals.

ELIGIBILITY:
Inclusion Criteria:

* ambulatory, post-menopausal women who would benefit from bisphosphonate treatment;
* >55 years of age;
* naive to bisphosphonate therapy, or lapsed bisphosphonate users >=6 months.

Exclusion Criteria:

* inability to stand or sit in an upright position for at least 60 minutes;
* hypersensitivity to bisphosphonates;
* treatment with other drugs affecting bone metabolism;
* history of major upper gastrointestinal disease.

Min Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 596 (Actual)
Dates: Start 2006-07; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Comparison of percentage of patients with persistence to >=10/12 administrations of Bonviva in feedback and no feedback group | 12 months

SECONDARY OUTCOMES:
Differences between groups in persistence | 6 months
QoL and patient satisfaction | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (168):
- France (168):
  - Agen
  - Aix-les-Bains
  - Albert
  - Amboise
  - Amiens
  - Andernos-les-Bains
  - Andrézieux-Bouthéon
  - Angers
  - Angoulême
  - Annecy
  - Antibes
  - Antony
  - Arcachon
  - Argeles
  - Arles
  - Armentières
  - Auch
  - Auray
  - Aurillac
  - Avignon
  - Avranches
  - Bayonne
  - Beaumont S/oise
  - Belfort
  - Besançon
  - Béziers
  - Billère
  - Blanquefort
  - Bolbec
  - Bordeaux
  - Brest
  - Bruz
  - Caen
  - Cagnes-sur-Mer
  - Cannes
  - Carpentras
  - Cavaillon
  - Cenon
  - Chalon-sur-Saône
  - Charenton-le-Pont
  - Chartres
  - Châlons-en-Champagne
  - Chelles
  - Chilly-Mazarin
  - Choisy-le-Roi
  - Clamart
  - Clermont-Ferrand
  - Clichy
  - Colmar
  - Cornebarrieu
  - Davézieux
  - Dax
  - Décines-Charpieu
  - Dijon
  - Dole
  - Fontaine
  - Fontenay S/bois
  - Gourdon
  - Granville
  - Grenoble
  - Hyères
  - Issy-les-Moulineaux
  - Istres
  - L'isle Sur Sorgue
  - L'Union
  - La Madeleine
  - La Roche-sur-Yon
  - La Rochelle
  - La Trinité
  - Lagny-sur-Marne
  - Landivisiau
  - Langon
  - Laval
  - Lavaur
  - Le Mans
  - Le Perreux-sur-Marne
  - Les Mureaux
  - Libourne
  - Lille
  - Limoges
  - Lisieux
  - Longwy
  - Loos
  - Lorient
  - Lyon
  - Maisons-Alfort
  - Mandelieu-la-Napoule
  - Marignane
  - Maromme
  - Marseille
  - Martigues
  - Meaux
  - Mennecy
  - Meylan
  - Mérignac
  - Millau
  - Miribel
  - Montbrisson
  - Montélimar
  - Montgeron
  - Montluçon
  - Montpellier
  - Mulhouse
  - Muret
  - Nancy
  - Nantes
  - Narbonne
  - Neuilly-sur-Seine
  - Nice
  - Nîmes
  - Nogent-le-Rotrou
  - Noisy-le-Sec
  - Oloron-Sainte-Marie
  - Orléans
  - Ormesson-sur-Marne
  - Orthez
  - Oyonnax
  - Pantin
  - Paris
  - Perpignan
  - Plan-de-Cuques
  - Poissy
  - Poitiers
  - Pont-à-Mousson
  - Puteaux
  - Quimper
  - Reims
  - Rennes
  - Rochefort
  - Ronchin
  - Roquebrune-Cap-Martin
  - Rouen
  - Rueil-Malmaison
  - Saint-Affrique
  - Saint-Brieuc
  - Saint-Doulchard
  - Saint-Etienne
  - Saint-Flour
  - Saint-Jacques-de-la-Lande
  - Saint-Lô
  - Saint-Mandé
  - Saint-Nazaire
  - Saint-Pierre-de-Coutances
  - Saint-Quentin
  - Sainte-Maxime
  - Saintes
  - Sarrebourg
  - Sartrouville
  - Sedan
  - Senlis
  - Sélestat
  - St-Malo
  - Strasbourg
  - Tassin-la-Demi-Lune
  - Thionville
  - Toulon
  - Toulouse
  - Tourcoing
  - Tournon-sur-Rhône
  - Tours
  - Valenciennes
  - Vandœuvre-lès-Nancy
  - Vence
  - Vernet-les-Bains
  - Vénissieux
  - Villeneuve-sur-Lot
  - Villeurbanne
  - Vincennes

REFERENCES:
- [Derived] Roux C, Giraudeau B, Rouanet S, Dubourg G, Perrodeau E, Ravaud P. Monitoring of bone turnover markers does not improve persistence with ibandronate treatment. Joint Bone Spine. 2012 Jul;79(4):389-92. doi: 10.1016/j.jbspin.2011.05.001. Epub 2011 Jun 23. PMID 21703900